CLINICAL TRIAL: NCT00483457
Title: Pilot Study of the Effects of Epidermal Growth Factor Receptor (EGFR) Inhibitors on the EGFR in Skin Lesions
Brief Title: Effects of Epidermal Growth Factor Receptor Inhibitor Therapy in the Skin of Cancer Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura W. Goff, MD, Assistant Professor of Medicine; Associate Director, Hematology/Oncology Fellowship Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC GI 0561; VU-VICC-GI-0561; VU-VICC-IRB-051020
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Solid Tumor
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Immunohistochemistry; Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: enzyme inhibitor therapy — enzyme inhibitor therapy
Genetic: protein expression analysis — protein expression analysis
Other: immunohistochemistry staining method — immunohistochemistry staining method
Other: laboratory biomarker analysis — laboratory biomarker analysis
Procedure: biopsy — biopsy

SUMMARY:
RATIONALE: Studying samples of tissue and blood in the laboratory from patients with cancer receiving epidermal growth factor receptor (EGFR) inhibitors may help doctors understand the effects of EGFR inhibitor therapy in the skin.

PURPOSE: This laboratory study is looking at the effects of EGFR inhibitors in the skin of cancer patients.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of EGFR inhibitors on the EGFR pathway in the skin of cancer patients prior to and after receiving EGFR inhibitors (i.e., tyrosine kinase inhibitors and monoclonal antibodies).
* Compare the effects of EGFR tyrosine kinase inhibitors vs monoclonal antibodies on the EGFR pathway in the skin of these patients.
* Compare changes in the EGFR pathway with grade of rash in these patients.
* Compare changes in EGFR pathway effectors in the skin with serum TGFα levels in these patients.

OUTLINE: This is a pilot study.

Patients undergo skin punch biopsies and blood sample collection at baseline, within 1 week of developing skin rash, and 6 weeks after beginning treatment. Samples are analyzed by immunohistochemistry and western blot for phosphorylated MAP kinase, AKT, and EGF levels and TGFα levels. Patients also complete diagrams to indicate locations of the rash once weekly during the first 6 weeks of treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a malignancy for which therapy on or off a clinical trial with an inhibitor of the EGFR pathway is under consideration

  * The therapy under consideration may be monotherapy or combined with other therapies as long as other therapies do not typically cause a rash

PATIENT CHARACTERISTICS:

* INR ≤ 3.0 (for patients receiving concurrent warfarin)
* No severe underlying skin disorder (e.g., toxic epidermal necrolysis or severe dermatitis) that would preclude study treatment
* No bleeding diatheses that would preclude safe biopsy
* No allergy to lidocaine or similar local anesthetics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients must be ≥ 18 years of age, have the diagnosis of a malignancy for which they are considering therapy with an inhibitor of the EGFR pathway, have no severe underlying skin disorder, must not have a bleeding diathesis that would preclude safe biopsy and patients on coumadin must not have an INR > 3.0 at time of biopsy.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Effects of EGFR inhibitors on the EGFR pathway in the skin prior to and after receiving EGFR inhibitors | baseline and at 6 weeks

SECONDARY OUTCOMES:
Comparison of the effects of EGFR tyrosine kinase inhibitors vs monoclonal antibodies on the EGFR pathway in the skin | at 6 weeks
Comparison of changes in the EGFR pathway with grade of rash | at 6 weeks
Comparison of changes in EGFR pathway effectors in the skin with serum TGFα levels as assessed by immunohistochemistry and western blot | at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goff, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States